CLINICAL TRIAL: NCT03371459
Title: A Randomized, Cumulative Dose, Open-label, 2-period Crossover, Multi-center Study to Assess the Safety, Efficacy, PK, and Extrapulmonary Pharmacodynamics (PD) of Cumulative Doses of Albuterol Sulfate Pressurized Inhalation Suspension (Hereafter Referred to as AS MDI) Compared to Cumulative Doses of Proventil® Hydrofluoroalkane (HFA; Hereafter Referred to as Proventil) as an Active Control in Subjects With Mild to Moderate Asthma (ASPEN)
Brief Title: Assessment of the Safety, Efficacy, PK, and Extrapulmonary Pharmacodynamics (PD) of Albuterol Sulfate Pressurized Inhalation Suspension (Hereafter Referred to as AS MDI) Compared to Proventil as an Active Control in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6930C00002
Record Dates: First submitted 2017-12-01; First posted 2017-12-13 (Actual); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AS MDI (Experimental): AS MDI 1+1+2+4+8 inhalations of 90 μg per inhalation
  Interventions: Drug: AS MDI
- Proventil (Active Comparator): Proventil 1+1+2+4+8 inhalations of 90 μg per inhalation
  Interventions: Drug: Proventil

INTERVENTIONS:
Drug: AS MDI — AS MDI 1+1+2+4+8 inhalations of 90 μg per inhalation
  Arms: AS MDI
Drug: Proventil — Proventil 1+1+2+4+8 inhalations of 90 μg per inhalation
  Arms: Proventil

SUMMARY:
This is a randomized, cumulative dose, open-label, 2-period crossover, multi-center study to assess the safety, efficacy, PK, and extrapulmonary PD of cumulative doses of AS MDI compared to cumulative doses of Proventil as an active control in subjects with mild to moderate asthma

DETAILED DESCRIPTION:
This is a randomized, cumulative dose, open-label, 2-period crossover, multi-center study to assess the safety, efficacy, PK, and extrapulmonary pharmacodynamics (PD) of cumulative doses of Albuterol Sulfate Pressurized Inhalation Suspension (hereafter referred to as AS MDI) compared to cumulative doses of Proventil® hydrofluoroalkane (HFA; hereafter referred to as Proventil) as an active control in subjects with mild to moderate asthma.

ELIGIBILITY:
Inclusion Criteria:

* Have stable (for 6 months) physician-diagnosed asthma with historical documentation of the diagnosis
* Must be receiving 1 of the following required inhaled asthma therapies listed below for at least the last 30 days; Only SABA, which is used as needed for rescue, or Low to medium doses of ICS (alone or in combination with LABA), used regularly as maintenance asthma therapy
* Demonstrate acceptable spirometry performance (ie, meet American Thoracic Society [ATS]/European Respiratory Society [ERS] acceptability/repeatability criteria
* Pre-bronchodilator FEV1 of ≥50 to <80% predicted normal value after withholding SABA ≥6 hours
* Confirmed FEV1 reversibility to Ventolin, defined as a post-Ventolin increase in FEV1 of ≥15%
* Only 2 reversibility testing attempts are allowed

Exclusion Criteria:

* Chronic obstructive pulmonary disease or other significant lung disease (eg, chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, or bronchopulmonary dysplasia)
* Oral corticosteroid use (any dose) within 6 weeks
* Received any marketed (eg, omalizumab, mepolizumab, reslizumab) or investigational biologic within 3 months or 5 half-lives, whichever is longer, or any other medication specifically prohibited by the protocol
* Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months (including all forms of tobacco, e-cigarettes [vaping], and marijuana)
* Life-threatening asthma as defined as any history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s)
* Historical or current evidence of a clinically significant disease
* Cancer not in complete remission for at least 5 years
* Hospitalized for psychiatric disorder or attempted suicide within 1 year
* Unable to abstain from protocol-defined prohibited medications during the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Winter Park, Florida
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Raleigh, North Carolina
  - Research Site, Medford, Oregon

REFERENCES:
- [Derived] Cappelletti C, Maes A, Rossman K, Gillen M, LaForce C, Kerwin EM, Reisner C. Dose-Ranging and Cumulative Dose Studies of Albuterol Sulfate MDI in Co-Suspension Delivery Technology (AS MDI; PT007) in Patients with Asthma: the ASPEN and ANTORA Trials. Clin Drug Investig. 2021 Jun;41(6):579-590. doi: 10.1007/s40261-021-01040-7. Epub 2021 Jun 4. PMID 34089147
- See also: Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14767&filename=PT007002_Redacted_Protocol_PDFA.pdf
- See also: Statistical Analysis Plan (SAP) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14767&filename=PT007002_Redacted_SAP_PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who met all screening and randomization requirements were eligible for rand to Tx Period, comprised of Visits 2 and 3 . Eligible subj were rand via IWRS to receive 2 cumulative-dose Tx's in one of 2 possible Tx sequences: AS MDI, given as 1+1+2+4+8 actuations of AS MDI 90 μg, Proventil, given as 1+1+2+4+8 actuations of Proventil 90 μg
Groups:
- Treatment Sequence A: AS MDI 90 ug then Proventil 90 ug
- Treatment Sequence B: Proventil 90 ug then AS MDI 90 ug
Period: Period 1
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0
Period: Washout
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 23 | 23
Completed | 23 | 22
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Period 2
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- mITT Population: The mITT Analysis Set is defined as a subset of the ITT Analysis Set including subjects who received treatment and had post-treatment efficacy data from both Treatment Periods. Data judged to be impacted by major protocol deviations are determined prior to database lock in a blinded fashion and excluded per the statistical protocol deviation plan. Statistical tabulations and analyses are by randomized treatment, but data obtained after subjects received an incorrect treatment are excluded from the affected periods
Arm/Group | mITT Population
Number analyzed (Participants) | 46
Age, Continuous [Least Squares Mean (Standard Deviation); unit: Years] — Population: mITT Population
  Years
    number analyzed (Participants) | 45
    (all) | 34.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: mITT Population
  Participants
    number analyzed (Participants) | 45
    Female | 22
    Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: mITT Population
  Participants
    number analyzed (Participants) | 45
    Hispanic or Latino | 7
    Not Hispanic or Latino | 38
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: mITT Population
  Participants
    number analyzed (Participants) | 45
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 11
    White | 34
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline-adjusted FEV1 30 Minutes After Each Cumulative Dose
Description: Forced expiratory volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation
Time Frame: At the two study treatment visits, FEV1 (forced expiratory volume in 1 second) will be measured prior to drug administration and 5 times, once at 30 minutes after each of the 5 doses
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Groups:
- AS MDI: AS MDI 90 μg 1+1+2+4+8 inhalations of 90 μg per inhalation
Arm/Group | AS MDI | Proventil
Number analyzed (Participants) | 45 | 45
Liter
  Dose 1 - 90 μg | 0.421 [0.300 to 0.543] | 0.488 [0.367 to 0.610]
  Cumulative Dose - 180 μg | 0.548 [0.432 to 0.665] | 0.586 [0.469 to 0.702]
  Cumulative Dose - 360 μg | 0.619 [0.502 to 0.737] | 0.647 [0.529 to 0.765]
  Cumulative Dose - 720 μg | 0.659 [0.544 to 0.775] | 0.690 [0.575 to 0.805]
  Cumulative Dose - 1440 μg | 0.721 [0.602 to 0.840] | 0.805 [0.686 to 0.925]

2. Secondary Outcome: Baseline-adjusted FEV1 AUC0-6 After the Last Cumulative Dose
Description: The baseline-adjusted FEV1 AUC0-6 is the area under the curve for change from baseline calculated using the trapezoidal rule and normalized by dividing the AUC by the length of follow up post the last cumulative dose (typically 6 hours) (spirometry will be obtained at 5, 15, 30, 45, 60, 120, 180, and 240 minutes post-dose) normalized for length of follow up).
Time Frame: Over 6 hours post dose on Day 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | AS MDI | Proventil
Number analyzed (Participants) | 45 | 45
Liter | 0.561 [0.448 to 0.674] | 0.602 [0.489 to 0.715]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed informed consent throughout the treatment period and up to 14 days following the last dose of study drug
Description: Serious Adverse Events were collected from the time the subject signed informed consent until study completion for a maximum of 44 days. This reporting time frame includes the screening period, the two active treatment periods, and the follow up period (i.e. 3-7 days after last dose of study drug).
Arm/Group | AS MDI | Proventil
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 8/45 | 10/46
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AS MDI (N=45) | Proventil (N=46)
Feeling Jittery (General disorders) | 3 (3) | 6 (6) — MedDRA
Tremor (Nervous system disorders) | 2 (2) | 2 (2) — MedDRA
Headache (Nervous system disorders) | 2 (2) | 0 (0) — MedDRA
Blood Potassium decreased (Investigations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT03371459/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03371459/SAP_001.pdf